CLINICAL TRIAL: NCT04376762
Title: Comparison of Fibrinogen Concentrate and Cryoprecipitate in Pediatric Cardiac Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Octapharma (Industry)
Responsible Party: Principal Investigator, Jacob Raphael, Professor UVA Department of Anesthesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSR180028-FC vs Cryo
Record Dates: First submitted 2020-02-26; First posted 2020-05-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pediatric HD; Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Fibrinogen; Injections; cryoprecipitate coagulum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fibrinogen Concentrate (Experimental): Fibrinogen Concentrate (dose: 70 mg/kg; intervention group). in-whom fibrinogen supplementation after separation from CPB is indicated, based on the presence of clinically-significant bleeding and documentation of low fibrinogen level on viscoelastic point-of-care testing (MCF < 10 mm on the FIBTEM assay of ROTEM).
  Interventions: Drug: Fibrinogen
- Cryoprecipitate (Active Comparator): . Cryoprecipitate (dose: 10 ml/kg; active control group) in-whom fibrinogen supplementation after separation from CPB is indicated, based on the presence of clinically-significant bleeding and documentation of low fibrinogen level on viscoelastic point-of-care testing (MCF < 10 mm on the FIBTEM assay of ROTEM).
  Interventions: Drug: Cryoprecipitate

INTERVENTIONS:
Drug: Fibrinogen — Fibrinogen Concentrate (Human) Injection [Fibryga] (dose: 70 mg/kg; intervention group). in-whom fibrinogen supplementation after separation from CPB is indicated, based on the presence of clinically-significant bleeding and documentation of low fibrinogen level on viscoelastic point-of-care testing (MCF < 10 mm on the FIBTEM assay of ROTEM).
  Other Names: Fibrinogen Concentrate (Human) Injection [Fibryga]
  Arms: Fibrinogen Concentrate
Drug: Cryoprecipitate — Cryoprecipitate group (dose: 10 ml/kg; active control group) in-whom fibrinogen supplementation after separation from CPB is indicated, based on the presence of clinically-significant bleeding and documentation of low fibrinogen level on viscoelastic point-of-care testing (MCF < 10 mm on the FIBTEM assay of ROTEM).
  Arms: Cryoprecipitate

SUMMARY:
The aim of the current pilot study proposal is to compare the use of the purified human fibrinogen concentrate (Fibryga®, Octapharma USA) to cryoprecipitate for the treatment of cardiopulmonary bypass (CPB)-associated bleeding in pediatric cardiac patients in whom fibrinogen supplementation is indicated.

The investigators' hypothesis is that fibrinogen concentrate will be as effective as cryoprecipitate in achieving adequate hemostasis after separation from CPB in pediatric cardiac surgery patients.

Study Design: this will be a single-center, prospective, randomized, active-control study in pediatric (24 months of age or younger) patients undergoing elective cardiac surgery with CPB (n=30) in-whom fibrinogen supplementation after separation from CPB is indicated, based on the presence of clinically-significant bleeding and documentation of low fibrinogen level on viscoelastic point-of-care testing (MCF < 10 mm on the FIBTEM assay of ROTEM). Informed consent will be obtained from a parent or a legal guardian prior to surgery and anesthesia. Once the need for fibrinogen supplementation is confirmed, study participants will be randomized into one of two treatment groups (n=15 in each group):

1. Cryoprecipitate group (dose: 10 ml/kg; active control group) or
2. Fibrinogen Concentrate group (dose: 70 mg/kg; intervention group). There will be no placebo group since withholding treatment is neither consistent with standard of care nor acceptable ethically. No other aspects of care will be modified. In the event that an additional dose of fibrinogen supplementation is required (bleeding with documented hypofibrinogenemia) cryoprecipitate will be administered to all study subjects (including those who received FC).

The results of this study will be used for publication as well as the first stage towards a significantly larger randomized multi-center trial (see below).

Based on the results of this pilot study the investigators plan to conduct a large multi-center, randomized active-control non-inferiority trial in the future, comparing the use of FC to cryoprecipitate in a much larger cohort of pediatric patients undergoing cardiac surgery with CPB. Ultimately, the results of this trial are likely to improve the care of pediatric cardiac surgical patients experiencing post-CPB bleeding, an under-studied yet high-risk patient population.

DETAILED DESCRIPTION:
Once the need for fibrinogen supplementation is confirmed, study participants will be randomized into one of two treatment groups (n=15 in each group):

1. Cryoprecipitate group (dose: 10 ml/kg; active control group) or
2. Fibrinogen Concentrate group (dose: 70 mg/kg; intervention group). There will be no placebo group since withholding treatment is neither consistent with standard of care nor acceptable ethically. No other aspects of care will be modified. In the event that an additional dose of fibrinogen supplementation is required (bleeding with documented hypofibrinogenemia) cryoprecipitate will be administered to all study subjects (including those who initially received FC).

Data to be obtained:

1. Demographic/preoperative data:

   * age in days/months (all participants to be 24 months of age or younger)
   * gender
   * weight
   * preoperative diagnosis
   * RACHS classification
   * surgery type & date (Norwood, arterial switch, truncus arteriosus, Glenn, anomalous pulmonary venous return, AV canal, tetralogy of Fallot, VSD closure, etc)
   * preoperative PT/INR/aPTT/hemoglobin level/ hematocrit/ platelet count/ WBC count/ fibrinogen level (Clauss method)
   * metabolic panel (sodium, BUN, creatinine, glucose, calcium, bicarbonate, Liver function tests)
2. Intra-operative Data:

   * CPB time & aortic cross clamp time
   * Use of hypothermic circulatory arrest (ice packs placed on the head)
   * ROTEM: Extem (CT/A10/A20/MCF) and Fibtem (A10/A20/MCF) at the following time points: baseline (after induction of anesthesia), 20 min prior to separation from CPB and 10 minutes after completion of fibrinogen concentrate/cryoprecipitate administration
   * Platelet count prior to separation from CPB
   * was ATIII administered? (thrombate)
   * Transfusion requirements: PRBC/Cell Saver/FFP/PLT/ cryoprecipitate - to be collected as number of units per each product, not volume. (for PLT - was it pooled PLT or single donor apheresis)
   * was rFVIIa given (factor seven, novoseven).
   * Need for ECMO support after separation trial from CPB
   * Was the chest left open?
3. Postoperative Data

   * PT/aPTT/INR/platelet count/ fibrinogen level/ Hgb level/HCT level on admission to the ICU
   * ROTEM parameters
   * Liver and kidney function tests on admission to the ICU
   * Bleeding (Chest drain output until 48 hours after surgery)
   * Need for additional transfusion (RBC/FFP/platelets/cryoprecipitate) until 7 days after surgery.
   * Factor VIIa administration
   * re-exploration for bleeding/tamponade (need for postoperative chest re-exploration or re- operation either in the ICU or in the OR due to excessive postoperative bleeding and/or cardiac tamponade)
   * Need for initiation of ECMO support in the ICU postoperatively
   * Duration of postoperative intubation
   * AKI (AKIN criteria)
   * Stroke/seizures > 24 hours post-operatively
   * Infection (sternal wound infection/mediastinitis/pneumonia/sepsis)
   * Thromboembolic complications (shunt thrombosis/DVT/PE)
   * ICU length of stay
   * Hospital length of stay
   * In hospital mortality

ELIGIBILITY:
Inclusion Criteria:

* pediatric (age 24 months or younger) patients undergoing elective cardiac surgery with CPB (n=30) in-whom fibrinogen supplementation after separation from CPB is indicated, based on the presence of clinically-significant bleeding and documentation of low fibrinogen level on viscoelastic point-of-care testing (MCF < 10 mm on the FIBTEM assay of ROTEM).

Exclusion Criteria:

* gestational age < 33 weeks at birth
* gestational age < 35 weeks on the day of surgery
* emergency surgery
* patient or parent history of coagulopathy/clotting abnormalities
* patient history of thrombophilia
* refusal to participate in the study,
* known severe allergic reaction/anaphylaxis to fibrinogen concentrate,
* administration of fibrinogen concentrate or cryoprecipitate in the 24 hours prior to surgery
* baseline fibrinogen level higher than 300 mg/dL (to avoid the risk of increasing the fibrinogen level above the normal upper level of 400 mg/dL)

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
A composite of the number of any allogeneic blood products (RBCs, plasma, platelets, cryoprecipitate) transfused from administration of the study medication until 48 hours after surgery | from immediately after the administration of the fibrinogen concentrate or cryoprecipitate through the first 48 hours after admission to the ICU/post anesthesia care unit
  comparison between study groups of the number of allogeneic blood products transfused (RBC, plasma, platelets, cryoprecipitate) from immediately after the administration of the study drug (fibrinogen concentrate or cryoprecipitate) until 48 hours since admission to the ICU

SECONDARY OUTCOMES:
Comparison of post CPB bleeding (in ml) between the study groups | from administration of fibrinogen concentrate or cryoprecipitate until 48 hours after primary postoperative admission to the ICU
  (intraoperatively = cell saver volume in ml; postoperatively = chest drain output in ml)
Comparison of the number RBC units transfused immediately after administration of the study medication and until postoperative day 7 | From immediately after study medication administration through postoperative day 7
  Comparison between the study groups of the number of RBC units transfused immediately after administration of the study medication (fibrinogen concentrate or cryoprecipitate) until postoperative day 7
Comparison of the number platelets units transfused immediately after administration of the study medication and until postoperative day 7 | From immediately after study medication administration through postoperative day 7
  Comparison between the study groups of the number of platelets units transfused immediately after administration of the study medication (fibrinogen concentrate or cryoprecipitate) until postoperative day 7
Comparison of the number plasma units transfused immediately after administration of the study medication and until postoperative day 7 | From immediately after study medication administration through postoperative day 7
  Comparison between the study groups of the number of plasma units transfused immediately after administration of the study medication (fibrinogen concentrate or cryoprecipitate) until postoperative day 7
Comparison of additional number cryoprecipitate units transfused immediately after administration of the study medication and until postoperative day 7 | From immediately after study medication administration through postoperative day 7
  Comparison between the study groups of the number of additional cryoprecipitate units transfused immediately after administration of the study medication (fibrinogen concentrate or cryoprecipitate) until postoperative day 7
Incidence of postoperative surgical chest re-exploration for excessive bleeding/cardiac tamponade | from admission to the ICU until postoperative day 7
  Comparison between study groups of the incidence of postoperative surgical chest re-exploration in the ICU/OR for excessive bleeding or cardiac tamponade
Incidence of the use of Factor VIIa for bleeding | from separation from CPB until 48 hours after surgery
  comparison of percent of patients requiring factor VIIa for bleeding (intraoperatively or postoperatively in the ICU between the study groups
In-hospital mortality | from admission to the ICU until 30 days after the operation/discharge from the hospital (whichever is earlier)
  comparison of the incidence of in-hospital mortality between the study groups
Post operative Acute Kidney injury (AKI) | from admission to the ICU until postoperative day 7
  comparison of the incidence of postoperative AKI between study groups. AKI will be assessed based on the Acute Kidney Injury Network (AKIN) classification (stages 0-3, with higher stage reflecting worse outcome)
Postoperative infection | rom admission to the ICU until 30 days after the operation/discharge from the hospital (whichever is earlier)
  comparison of the incidence of pneumonia, sternal wound infection, mediastinitis, sepsis between study groups
percent of patients with postoperative neurological injury | from admission to the ICU until POD 7
  Comparison between study groups of the percent of patients with seizures/stroke that occur after surgery
Intubation time | from admission to the ICU until 30 days after surgery or discharge from the ICU (whichever is earlier)
  comparison of the time to extubation from the completion of surgery until extubation in the ICU between the study groups
postoperative thromboembolic event | from admission to the ICU until 7 days postoperatively
  comparison of the incidence of DVT/PE/shunt thrombosis between the study groups
ICU length of stay | from admission to the ICU after surgery until 90 days after surgery or discharge from the ICU (whichever occurs earlier)
  comparison of the postoperative time period spent in the ICU
Hospital length of stay | from admission to the ICU postoperatively until postoperative day 90 or discharge from the hospital (whichever occurs earlier)
  comparison between the study groups of the time in the hospital from admission to the ICU postoperatively until discharge from the hospital

OTHER OUTCOMES:
Percent of patients requiring postoperative Extra Corporeal Membrane Oxygenation (ECMO) support | from separation from CPB until postoperative day 30 (or discharge from the hospital (whichever occurs earlier)
  comparison between the groups of the incidence of the need for postoperative circulatory support with ECMO

CONTACTS AND LOCATIONS:
Overall Officials: Keita Ikeda, MD, Study Director — UVA Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hvas AM, Andreasen JB, Christiansen K, Ravn HB. Ex-vivo response to blood products and haemostatic agents after paediatric cardiac surgery. Blood Coagul Fibrinolysis. 2013 Sep;24(6):587-92. doi: 10.1097/MBC.0b013e32836029d2. PMID 23571685
- [Background] Galas FR, de Almeida JP, Fukushima JT, Vincent JL, Osawa EA, Zeferino S, Camara L, Guimaraes VA, Jatene MB, Hajjar LA. Hemostatic effects of fibrinogen concentrate compared with cryoprecipitate in children after cardiac surgery: a randomized pilot trial. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1647-55. doi: 10.1016/j.jtcvs.2014.04.029. Epub 2014 Apr 18. PMID 24951020
- [Background] Haas T, Spielmann N, Restin T, Seifert B, Henze G, Obwegeser J, Min K, Jeszenszky D, Weiss M, Schmugge M. Higher fibrinogen concentrations for reduction of transfusion requirements during major paediatric surgery: A prospective randomised controlled trial. Br J Anaesth. 2015 Aug;115(2):234-43. doi: 10.1093/bja/aev136. Epub 2015 May 15. PMID 25982134
- [Background] Haas T, Cushing MM, Asmis LM. Comparison of the efficacy of two human fibrinogen concentrates to treat dilutional coagulopathy in vitro. Scand J Clin Lab Invest. 2018 May;78(3):230-235. doi: 10.1080/00365513.2018.1437645. Epub 2018 Feb 15. PMID 29446989
- [Background] Ranucci M, Baryshnikova E, Crapelli GB, Rahe-Meyer N, Menicanti L, Frigiola A; Surgical Clinical Outcome REsearch (SCORE) Group. Randomized, double-blinded, placebo-controlled trial of fibrinogen concentrate supplementation after complex cardiac surgery. J Am Heart Assoc. 2015 Jun 2;4(6):e002066. doi: 10.1161/JAHA.115.002066. PMID 26037084
- [Background] Fassl J, Lurati Buse G, Filipovic M, Reuthebuch O, Hampl K, Seeberger MD, Bolliger D. Perioperative administration of fibrinogen does not increase adverse cardiac and thromboembolic events after cardiac surgery. Br J Anaesth. 2015 Feb;114(2):225-34. doi: 10.1093/bja/aeu364. Epub 2014 Oct 16. PMID 25324348